CLINICAL TRIAL: NCT00322452
Title: Open Label, Randomised, Parallel Group, Multicentre, Ph III Study To Assess Efficacy, Safety & Tolerability Of Gefitinib (IRESSA™) Versus Carboplatin/Paclitaxel DC As 1st-Line Treatment In Selected Patients With Stage IIIB / IV NSCLC In Asia
Brief Title: First Line IRESSA™ Versus Carboplatin/Paclitaxel in Asia
Acronym: IPASS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D791AC00007; Iressa Pan Asian Study (IPASS)
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Results first posted 2010-05-17 (Estimated); Last update posted 2013-11-07 (Estimated); Status verified 2013-10

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; Gefitinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Carboplatin; Paclitaxel

ARMS (2):
- 1 (Experimental): gefitinib
  Interventions: Drug: Gefitinib
- 2 (Active Comparator): Carboplatin/Paclitaxel
  Interventions: Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Gefitinib — oral tablet
  Other Names: Iressa; ZD1839
  Arms: 1
Drug: Carboplatin — IV
  Arms: 2
Drug: Paclitaxel — IV
  Arms: 2

SUMMARY:
The purpose of this study is to compare gefitinib with carboplatin / paclitaxel doublet chemotherapy given as first line treatment in terms of progression free survival in selected NSCLC patients with the objective of demonstrating non-inferiority.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced Stage IIIB not amenable to local therapy or Stage IV (metastatic) NSCLC with adenocarcinoma histology.
* Never smokers or light ex-smokers.(ceased smoking at least 15 years before Day 1 of study treatment and 10 pack-years or fewer)

Exclusion Criteria:

* Had prior chemotherapy, biological (including targeted therapies such as EGFR and vascular epidermal growth factor (VEGF) inhibitors) or immunological therapy.
* Pre-existing idiopathic pulmonary fibrosis evidence by CT scan at baseline.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1329 (Actual)
Dates: Start 2006-03; Primary Completion 2008-04 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Armour, MD, Study Director — AstraZeneca
Locations (56):
- China (10):
  - Research Site, Fuzhou, Fujian
  - Research Site, Guangzhou, Guangdong
  - Research Site, Wuhan, Hubei
  - Research Site, Nanjing, Jiangsu
  - Research Site, Dalian, Liaoning
  - Research Site, Chongqing, Sichuan
  - Research Site, Beijing
  - Research Site, Chengdu
  - Research Site, Hangzhou
  - Research Site, Shanghai
- Research Site, Hong Kong, Hong Kong
- Indonesia (6):
  - Research Site, Semarang, Central Java
  - Research Site, Malang, East Java
  - Research Site, Jakarta
  - Research Site, Solo
  - Research Site, Surabaya
  - Research Site, Yogyakarta
- Japan (22):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Okazaki, Aichi-ken
  - Research Site, Kashiwa, Chiba
  - Research Site, Matsuyama, Ehime
  - Research Site, Fukuoka, Fukuoka
  - Research Site, Sapporo, Hokkaido
  - Research Site, Akashi, Hyōgo
  - Research Site, Kobe, Hyōgo
  - Research Site, Kanazawa, Ishikawa-ken
  - Research Site, Yokohama, Kanagawa
  - Research Site, Kumamoto, Kumamoto
  - Research Site, Ōmura, Nagasaki
  - Research Site, Okayama, Okayama-ken
  - Research Site, Izumisano, Osaka
  - Research Site, Osaka, Osaka
  - Research Site, Sakai, Osaka
  - Research Site, Sayama, Osaka
  - Research Site, Sunto-gun, Shizuoka
  - Research Site, Bunkyo-ku, Tokyo
  - Research Site, Koto-ku, Tokyo
  - Research Site, Shinjuku, Tokyo
  - Research Site, Ube, Yamaguchi
- Malaysia (5):
  - Research Site, Kota Kinabalu, Sabah
  - Research Site, George Town
  - Research Site, Kampung Baharu Nilai
  - Research Site, Kuala Lumpur
  - Research Site, Petaling Jaya
- Philippines (3):
  - Research Site, Cebu City
  - Research Site, Manila
  - Research Site, Quezon City
- Research Site, Singapore, Singapore
- Taiwan (4):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Khon Kaen
  - Research Site, Songkhla

REFERENCES:
- [Derived] Nagase M, Aksenov S, Yan H, Dunyak J, Al-Huniti N. Modeling Tumor Growth and Treatment Resistance Dynamics Characterizes Different Response to Gefitinib or Chemotherapy in Non-Small Cell Lung Cancer. CPT Pharmacometrics Syst Pharmacol. 2020 Mar;9(3):143-152. doi: 10.1002/psp4.12490. Epub 2020 Feb 7. PMID 31920008
- [Derived] Wu YL, Saijo N, Thongprasert S, Yang JC, Han B, Margono B, Chewaskulyong B, Sunpaweravong P, Ohe Y, Ichinose Y, Yang JJ, Mok TS, Young H, Haddad V, Rukazenkov Y, Fukuoka M. Efficacy according to blind independent central review: Post-hoc analyses from the phase III, randomized, multicenter, IPASS study of first-line gefitinib versus carboplatin/paclitaxel in Asian patients with EGFR mutation-positive advanced NSCLC. Lung Cancer. 2017 Feb;104:119-125. doi: 10.1016/j.lungcan.2016.11.022. Epub 2016 Nov 30. PMID 28212993
- [Derived] Yang JC, Wu YL, Chan V, Kurnianda J, Nakagawa K, Saijo N, Fukuoka M, McWalter G, McCormack R, Mok TS. Epidermal growth factor receptor mutation analysis in previously unanalyzed histology samples and cytology samples from the phase III Iressa Pan-ASia Study (IPASS). Lung Cancer. 2014 Feb;83(2):174-81. doi: 10.1016/j.lungcan.2013.11.021. Epub 2013 Dec 1. PMID 24361280
- [Derived] Wu YL, Fukuoka M, Mok TS, Saijo N, Thongprasert S, Yang JC, Chu DT, Yang JJ, Rukazenkov Y. Tumor response and health-related quality of life in clinically selected patients from Asia with advanced non-small-cell lung cancer treated with first-line gefitinib: post hoc analyses from the IPASS study. Lung Cancer. 2013 Aug;81(2):280-7. doi: 10.1016/j.lungcan.2013.03.004. Epub 2013 Mar 26. PMID 23540718
- [Derived] Wu YL, Chu DT, Han B, Liu X, Zhang L, Zhou C, Liao M, Mok T, Jiang H, Duffield E, Fukuoka M. Phase III, randomized, open-label, first-line study in Asia of gefitinib versus carboplatin/paclitaxel in clinically selected patients with advanced non-small-cell lung cancer: evaluation of patients recruited from mainland China. Asia Pac J Clin Oncol. 2012 Sep;8(3):232-43. doi: 10.1111/j.1743-7563.2012.01518.x. Epub 2012 Apr 23. PMID 22897752
- [Derived] Mok TS, Wu YL, Thongprasert S, Yang CH, Chu DT, Saijo N, Sunpaweravong P, Han B, Margono B, Ichinose Y, Nishiwaki Y, Ohe Y, Yang JJ, Chewaskulyong B, Jiang H, Duffield EL, Watkins CL, Armour AA, Fukuoka M. Gefitinib or carboplatin-paclitaxel in pulmonary adenocarcinoma. N Engl J Med. 2009 Sep 3;361(10):947-57. doi: 10.1056/NEJMoa0810699. Epub 2009 Aug 19. PMID 19692680

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Males or females that had never smoked or were light ex-smokers, who had Stage IIIB or Stage IV adenocarcinoma of the lung and had not received any previous chemotherapy excluding non-platinum based adjuvant chemotherapy were randomised between 30 March 2006 and 9 October 2007. The study was carried out in Asian countries (including Japan & China).
Pre-assignment Details: 112 patients (out of 1329) failed screening and were not randomized, the majority of patients who failed screening did not comply with inclusion / exclusion criteria. Other reasons were: patient withdrew informed consent; patient lost to follow up. One patient was not randomized for 'other' (non-specified) reason.
Groups:
- Gefitinib: Gefitinib 250mg daily
- Carboplatin/Paclitaxel: Carboplatin AUC 5.0 or 6.0 and Paclitaxel 200 mg/m^2 doublet chemotherapy every 3 weeks
Period: Overall Study
Arm/Group | Gefitinib | Carboplatin/Paclitaxel
Started | 609 (Number of patients randomized) | 608 (Number of patients randomized)
Completed | 362 (Patients still in study at PFS Data Cut Off (14 April 2008), 97 remained at OS DCO (14 June 2010)) | 332 (Patients still in study at PFS Data Cut Off (14 April 2008), 84 remained at OS DCO (14 June 2010))
Not Completed | 247 | 276
Not completed — Eligibility criteria not fulfilled | 0 | 1
Not completed — Lost to Follow-up | 5 | 2
Not completed — Withdrawal by Subject | 19 | 46
Not completed — Death | 223 | 227

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gefitinib | Carboplatin/Paclitaxel | Total
Number analyzed (Participants) | 609 | 608 | 1217
Age Continuous [Median (Full Range); unit: Years] | 57 [24 to 84] | 57 [25 to 84] | 57 [24 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 484 | 481 | 965
  Male | 125 | 127 | 252
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 3 | 1 | 4
  Oriental | 603 | 606 | 1209
  Other | 3 | 1 | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian (other than Chinese or Japanese) | 179 | 184 | 363
  Chinese | 314 | 304 | 618
  Japanese | 114 | 119 | 233
  Other | 2 | 1 | 3
Smoking history [Number; unit: Participants]
  Never Smoker | 571 | 569 | 1140
  Light ex-smoker | 37 | 38 | 75
  Ex-smoker (non-light) | 1 | 1 | 2
WHO performance status [Number; unit: Participants]
  0 (normal activity) | 157 | 161 | 318
  1 (restricted activity) | 391 | 382 | 773
  2 (in bed =< 50% of the time) | 61 | 65 | 126

OUTCOME MEASURES:

1. Primary Outcome: Median Progression Free Survival (PFS) in Months
Description: PFS was defined as the interval from the date of randomization to the date of objective disease progression (as per RECIST) or the date of death (from any cause) in the absence of objective disease progression. The median PFS in months is presented here.
Time Frame: Tumour assessments as per RECIST were performed at baseline and then every 42 days ± 7 days from randomization until data cut off (14th April 2008).
Population: Analysis was carried out on Intention-to-treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gefitinib | Carboplatin/Paclitaxel
Number analyzed (Participants) | 609 | 608
Months | 5.7 [5.4 to 6.8] | 5.8 [5.6 to 6.4]

2. Secondary Outcome: Median Overall Survival (OS) in Months at OS Data Cut Off (14th June 2010)
Description: Overall Survival was assessed via calculation of the time to death due to any cause. If a participant was known to have died, the time to death was defined as the time from the date of randomization to the date of death. Otherwise, a participant was censored at the last date they were known to be alive. Median Overall Survival in months is presented here.
Time Frame: Following the PFS DCO on 14th April 2008 information on survival status was collected every 8 weeks.
Population: Analysis was carried out on Intention-to-treat (ITT) population.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Gefitinib | Carboplatin/Paclitaxel
Number analyzed (Participants) | 609 | 608
Months | 18.8 [17.3 to 20.4] | 17.4 [16.2 to 18.7]

3. Secondary Outcome: Objective Tumour Response Rate According to RECIST
Description: Number of participants with an objective response. An objective response (OR) was defined as a patient having a best overall response of either complete response (CR) or partial response (PR) according to RECIST, confirmed at least 28 days following the date of the initial response.
Time Frame: as for outcome 1
Population: Analysis was carried out on Intention-to-treat (ITT) population.
Measure: Number; unit: Participants
Arm/Group | Gefitinib | Carboplatin/Paclitaxel
Number analyzed (Participants) | 609 | 608
Participants | 262 | 196

4. Secondary Outcome: Common Toxicity Criteria (CTC) Grade 3, 4, or 5 Neutropenia
Description: Number of patients with a neutropenia event, identified from the lab data as a worsening in absolute neutrophil count from baseline to a CTC grade 3 or above which Based on the evaluable-for-safety population, which included all patients who received at least 1 dose of study medication (gefitinib, or carboplatin or paclitaxel).
Time Frame: Includes events that occurred whilst a patient was receiving first-line randomized treatment: defined as date of first dose to date of last dose +1 day for gefitinib, and date of first infusion to date of last infusion + 21 days for carboplatin/paclitaxel
Population: Analysis was carried out on the Evaluable-for-safety (EFS) population. The EFS population is a subset of the ITT population which includes all patients who received at least 1 dose of study medication (gefitinib, or carboplatin or paclitaxel).
Measure: Number; unit: Participants
Arm/Group | Gefitinib | Carboplatin/Paclitaxel
Number analyzed (Participants) | 607 | 589
Participants | 4 | 385

5. Secondary Outcome: Common Toxicity Criteria (CTC) Grade 3, 4, or 5 Thrombocytopenia
Description: Number of patients with a thromboctyopenia event, identified from the lab data as a worsening in platelet count from baseline to a CTC grade 3 or above. Based on the evaluable-for-safety population, which included all patients who received at least 1 dose of study medication (gefitinib, or carboplatin or paclitaxel).
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Gefitinib | Carboplatin/Paclitaxel
Number analyzed (Participants) | 607 | 589
Participants | 5 | 29

6. Secondary Outcome: Common Toxicity Criteria (CTC) Grade 3, 4, or 5 Leukopenia
Description: Number of patients with a leukopenia event, identified from the lab data as a worsening in white blood cell count from baseline to a CTC grade 3 or above. Based on the evaluable for-safety-population, which included all patients who received at least 1 dose of study medication (gefitinib, or carboplatin or paclitaxel).
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Gefitinib | Carboplatin/Paclitaxel
Number analyzed (Participants) | 607 | 589
Participants | 1 | 202

7. Secondary Outcome: Common Toxicity Criteria (CTC) Grade 3, 4, or 5 Anaemia
Description: Number of patients with an anaemia event, identified from the lab data as a worsening in haemoglobin from baseline to a CTC grade 3 or above. Based on the evaluable-for-safety population, which included all patients who received at least 1 dose of study medication (gefitinib, or carboplatin or paclitaxel).
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Gefitinib | Carboplatin/Paclitaxel
Number analyzed (Participants) | 607 | 589
Participants | 11 | 56

8. Secondary Outcome: Neurotoxicity
Description: Number of patients with a neurotoxicity event. Based on the evaluable-for-safety population, which included all patients who received at least 1 dose of study medication (gefitinib, or carboplatin or paclitaxel)
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Gefitinib | Carboplatin/Paclitaxel
Number analyzed (Participants) | 607 | 589
Participants | 30 | 411

9. Secondary Outcome: Rashes/Acnes
Description: Number of patients with a rashes/acnes event. Based on the evaluable-for-safety population, which included all patients who received at least 1 dose of study medication (gefitinib, or carboplatin or paclitaxel)
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Gefitinib | Carboplatin/Paclitaxel
Number analyzed (Participants) | 607 | 589
Participants | 398 | 132

10. Secondary Outcome: Diarrhoea
Description: Number of patients with a diarrhoea event. Based on the evaluable-for-safety population, which included all patients who received at least 1 dose of study medication (gefitinib, or carboplatin or paclitaxel)
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Gefitinib | Carboplatin/Paclitaxel
Number analyzed (Participants) | 607 | 589
Participants | 274 | 128

11. Secondary Outcome: Nausea
Description: Number of patients with a nausea event. Based on the evaluable for-safety-population, which included all patients who received at least 1 dose of study medication (gefitinib, or carboplatin or paclitaxel)
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Gefitinib | Carboplatin/Paclitaxel
Number analyzed (Participants) | 607 | 589
Participants | 74 | 260

12. Secondary Outcome: Vomiting
Description: Number of patients with a vomiting event. Based on the evaluable-for-safety population, which included all patients who received at least 1 dose of study medication (gefitinib, or carboplatin or paclitaxel)
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Gefitinib | Carboplatin/Paclitaxel
Number analyzed (Participants) | 607 | 589
Participants | 59 | 193

13. Secondary Outcome: Common Toxicity Criteria (CTC) Grade 3, 4, or 5 Liver Transaminases
Description: Number of patients with an elevated liver transaminase event, identified from the lab data as a worsening in ALT or AST from baseline to a CTC grade 3 or above. Based on the evaluable-for-safety population, which included all patients who received at least 1 dose of study medication (gefitinib, or carboplatin or paclitaxel).
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Number; unit: Participants
Arm/Group | Gefitinib | Carboplatin/Paclitaxel
Number analyzed (Participants) | 607 | 589
Participants | 57 | 6

14. Secondary Outcome: Quality of Life (QoL) as Measured by the Total Score of the Functional Assessment of Cancer Therapy - Lung Cancer (FACT-L) Questionnaire
Description: Number of patients improving: a patient was described as improved if they had 2 visits (at least 21 days apart) where there was an increase in FACT-L score (from baseline) of 6 or more, and there were no intervening visits showing a decrease from baseline of 6 or more. Includes all patients with QoL data at baseline & at least 1 post-baseline visit
Time Frame: FACT-L data were collected at baseline, week 1, every 3 weeks (from baseline) until day 127, then every 42 days until the patient was confirmed as having objectively progressed (via RECIST), and at treatment discontinuation.
Population: Analysis was carried out on the Evaluable-for-QoL (EFQ) population. The EFQ population is a subset of the ITT population containing patients with an evaluable baseline QoL assessment and at least 1 evaluable post-baseline QoL assessment.
Measure: Number; unit: Participants
Arm/Group | Gefitinib | Carboplatin/Paclitaxel
Number analyzed (Participants) | 590 | 561
Participants | 283 | 229

15. Secondary Outcome: Quality of Life (QoL) as Measured by the Trial Outcome Index (TOI) of the Functional Assessment of Cancer Therapy - Lung Cancer (FACT-L) Questionnaire
Description: Number of patients improving: a patient was described as improved if they had 2 visits (at least 21 days apart) where there was an increase in TOI score (from baseline) of 6 or more, and there were no intervening visits showing a decrease from baseline of 6 or more. Includes all patients with QoL data at baseline & at least 1 post-baseline visit
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Number; unit: Participants
Arm/Group | Gefitinib | Carboplatin/Paclitaxel
Number analyzed (Participants) | 590 | 561
Participants | 274 | 184

16. Secondary Outcome: Symptom Improvement as Measured by the Lung Cancer Subscale (LCS) of the FACT-L Questionnaire
Description: Number of patients improving: a patient was described as improved if they had 2 visits (at least 21 days apart) where there was an increase in LCS score (from baseline) of 2 or more, and there were no intervening visits showing a decrease from baseline of 2 or more. Includes all patients with QoL data at baseline & at least 1 post-baseline visit
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Number; unit: Participants
Arm/Group | Gefitinib | Carboplatin/Paclitaxel
Number analyzed (Participants) | 590 | 561
Participants | 304 | 272

ADVERSE EVENTS:
Arm/Group | Gefitinib | Carboplatin/Paclitaxel
Serious Adverse Events (participants affected / at risk) | 110/607 | 92/589
Other Adverse Events (participants affected / at risk) | 574 | 573
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gefitinib (N=607) | Carboplatin/Paclitaxel (N=589)
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 1 | 1
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 0
Altered State Of Consciousness (Nervous system disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 5
Anaphylactic Shock (Immune system disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 1 | 1
Angle Closure Glaucoma (Eye disorders) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 0
Bone Marrow Failure (Blood and lymphatic system disorders) | 1 | 0
Brain Herniation (Injury, poisoning and procedural complications) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Calculus Urinary (Renal and urinary disorders) | 2 | 0
Cardiac Arrest (Cardiac disorders) | 0 | 1
Cardiac Failure (Cardiac disorders) | 1 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Cerebral Artery Embolism (Nervous system disorders) | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 2 | 0
Chest Pain (General disorders) | 3 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 1 | 1
Deep Vein Thrombosis (Vascular disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Depressed Level Of Consciousness (Nervous system disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Dizziness (Nervous system disorders) | 2 | 2
Drug Hypersensitivity (Immune system disorders) | 1 | 3
Duodenitis (Gastrointestinal disorders) | 0 | 1
Dysfunctional Uterine Bleeding (Reproductive system and breast disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Embolism (Vascular disorders) | 0 | 1
Encephalitis (Nervous system disorders) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 0
Fatigue (General disorders) | 0 | 2
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastric Ulcer Perforation (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 | 2
Haematuria (Renal and urinary disorders) | 1 | 0
Haemoglobin Decreased (Investigations) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 1 | 0
Hepatic Failure (Hepatobiliary disorders) | 1 | 0
Hepatic Function Abnormal (Hepatobiliary disorders) | 4 | 1
Herpes Zoster (Infections and infestations) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 1
Hypotension (Vascular disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Iiird Nerve Paralysis (Nervous system disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Ischaemic Stroke (Nervous system disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Lacunar Infarction (Nervous system disorders) | 1 | 0
Laryngeal Granuloma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 1
Lung Infection (Infections and infestations) | 0 | 1
Malaise (General disorders) | 0 | 2
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myocardial Infarction (Cardiac disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 10
Neutrophil Count Decreased (Investigations) | 0 | 2
Oral Intake Reduced (Metabolism and nutrition disorders) | 0 | 1
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain (General disorders) | 0 | 1
Parotitis (Infections and infestations) | 0 | 1
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 | 2
Pericardial Effusion (Cardiac disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Infections and infestations) | 9 | 9
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pseudomonal Sepsis (Infections and infestations) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pupils Unequal (Eye disorders) | 1 | 0
Pyothorax (Infections and infestations) | 2 | 0
Pyrexia (General disorders) | 3 | 2
Radius Fracture (Injury, poisoning and procedural complications) | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 1 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Sciatica (Nervous system disorders) | 1 | 0
Sepsis (Infections and infestations) | 2 | 0
Septic Shock (Infections and infestations) | 0 | 3
Sinus Bradycardia (Cardiac disorders) | 1 | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 | 0
Syncope Vasovagal (Nervous system disorders) | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Ventricular Tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Gefitinib | Carboplatin/Paclitaxel
Acne (Skin and subcutaneous tissue disorders) | 66/607 | 4/589
Alanine Aminotransferase Increased (Investigations) | 61/607 | 31/589
Alopecia (Skin and subcutaneous tissue disorders) | 42/607 | 343/589
Anaemia (Blood and lymphatic system disorders) | 36/607 | 146/589
Anorexia (Metabolism and nutrition disorders) | 92/607 | 232/589
Arthralgia (Musculoskeletal and connective tissue disorders) | 22/607 | 112/589
Aspartate Aminotransferase Increased (Investigations) | 52/607 | 19/589
Back Pain (Musculoskeletal and connective tissue disorders) | 32/607 | 26/589
Constipation (Gastrointestinal disorders) | 47/607 | 170/589
Cough (Respiratory, thoracic and mediastinal disorders) | 53/607 | 62/589
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 35/607 | 2/589
Diarrhoea (Gastrointestinal disorders) | 273/607 | 127/589
Dizziness (Nervous system disorders) | 31/607 | 35/589
Dry Skin (Skin and subcutaneous tissue disorders) | 144/607 | 17/589
Dyspepsia (Gastrointestinal disorders) | 32/607 | 26/589
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 35/607 | 49/589
Fatigue (General disorders) | 72/607 | 217/589
Haemoglobin Decreased (Investigations) | 1/607 | 30/589
Headache (Nervous system disorders) | 39/607 | 43/589
Hepatic Function Abnormal (Hepatobiliary disorders) | 48/607 | 23/589
Hypoaesthesia (Nervous system disorders) | 7/607 | 153/589
Hypokalaemia (Metabolism and nutrition disorders) | 20/607 | 30/589
Insomnia (Psychiatric disorders) | 72/607 | 107/589
Leukopenia (Blood and lymphatic system disorders) | 5/607 | 146/589
Myalgia (Musculoskeletal and connective tissue disorders) | 24/607 | 186/589
Nasopharyngitis (Infections and infestations) | 52/607 | 22/589
Nausea (Gastrointestinal disorders) | 74/607 | 259/589
Neuropathy Peripheral (Nervous system disorders) | 5/607 | 97/589
Neutropenia (Blood and lymphatic system disorders) | 3/607 | 218/589
Neutrophil Count Decreased (Investigations) | 0/607 | 39/589
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 24/607 | 40/589
Paraesthesia (Nervous system disorders) | 8/607 | 30/589
Paronychia (Infections and infestations) | 82/607 | 0/589
Peripheral Sensory Neuropathy (Nervous system disorders) | 9/607 | 141/589
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 36/607 | 28/589
Pruritus (Skin and subcutaneous tissue disorders) | 103/607 | 69/589
Pyrexia (General disorders) | 38/607 | 56/589
Rash (Skin and subcutaneous tissue disorders) | 308/607 | 120/589
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 31/607 | 1/589
Stomatitis (Gastrointestinal disorders) | 78/607 | 42/589
Thrombocytopenia (Blood and lymphatic system disorders) | 7/607 | 70/589
Upper Respiratory Tract Infection (Infections and infestations) | 34/607 | 23/589
Vomiting (Gastrointestinal disorders) | 58/607 | 190/589
White Blood Cell Count Decreased (Investigations) | 3/607 | 52/589

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator (PI) agrees to collaborate on the contents and formation of any publication and to pay due consideration to comments and opinions offered. AstraZeneca have 30 days for final manuscript review and may require that submission for publication be delayed in order to file patent applications.